CLINICAL TRIAL: NCT06159257
Title: Evaluation of the Physiological Stability Variability and Robustness of NIS4,a Serum Biomarker for the Diagnosis of Non-alcoholic Steaohepatitis
Brief Title: Evaluation of the Physiological Stability Variability and Robustness of NIS4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NASH
Record Dates: First submitted 2023-11-17; First posted 2023-12-06 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Evaluate the Physiological Stability of NIS4 Biomarker Between the Fed and Fasting State in Patients With the Target Condition (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steatohepatitis (NASH) (Other)
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Whenever possible, samples will be collected by the nurse in the patient's home, according to the study visit schedule. However, if this is not possible, patients will be asked to come in for sample collection at another mutually convenient time at the CERBA ALLIANCE LABORATORY closest to the patient's address.
  Venous blood will be drawn on each visit.

SUMMARY:
Patients at higher risk of progression to cirrhosis and clinical deleterious outcomes are those that have a high grade of necroinflammation together with significant fibrosis. This defines a level of disease severity which is called "at-risk NASH". Currently registrational trials for NASH include only patients with at-risk NASH so it is predictable that when a drug will be approved for NASH it will be in patients with at-risk NASH. It is therefore important to be able to diagnose non-invasively patients with at-risk NASH. Also, the use of NIS4 in clinical trials or in the clinic has the potential to significantly reduce unnecessary liver biopsies by identifying patients with a lower risk of disease progression. GENFIT, a late-stage biopharmaceutical company dedicated to improving the lives of patients with metabolic and chronic liver diseases, is developing an in vitro diagnostic test for at-risk NASH. The test is calledNIS4™ and integrates four independent biomarkers - miR-34a-5p, A2M, YKL-40 and HbA1c. The output is a score from 0 to 1 with threshold values that identify patients at low risk and high risk of at-risk NASH with intermediate values representing indeterminate results. The objective of the program is to complete the development of the predictive and usable NIS4 score and to evaluate the impact of fasting or not fasting on the physiological stability, variability and robustness of circulating biomarkers for the diagnosis of non-alcoholic steatohepatitis over a 30-day period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented steatohepatitis (NASH) with at least minimal (grade 1) hepatocyte ballooning and inflammation on a biopsy performed in the past year.
* OR, if a biopsy is not available:

  1. Presence of metabolic risk factors (see below) AND
  2. Documentation of steatosis on imaging (hepatic ultrasound, CT scan or MRI) AND
  3. Increased ALT >30 IU/L OR liver stiffness >5 kPa on Fibroscan
* Metabolically stable condition, in particular no weight change >5% in the past 6 months, anticipated stable diabetic therapy during the study period
* No other identifiable cause of liver disease
* Patients affiliated to French social security.
* Written informed consent signed by the patient

Exclusion Criteria:

* Patient with Hepatitis B or C.
* Presence of any other form of chronic liver disease
* Average alcohol consumption greater than 20 g/day for females and 30 g/day for males in the preceding 6 months or history of sustained excessive consumption of alcohol in past 5 years.
* Severely uncontrolled diabetes (HbA1c>9.5%)
* Recent (within 12 months) or concomitant use of agents known to cause hepatic steatosis (long-term systemic corticosteroids [>10 days], amiodarone, methotrexate, tamoxifen, tetracycline, high dose oestrogens, valproic acid).
* Recent (within 3 months) change in dose/regimen or introduction of Vitamin E (at a dose ≥400 IU/day), betaine, s-adenosyl methionine, ursodeoxycholic acid, silymarin or pentoxifylline.
* HIV infection.
* Person not fasted 12 hours (T10, T12, D0).
* Substantial diet modification in the 4 months prior to inclusion.
* Patients judged by the investigator to be unsuitable for inclusion in the study (e.g., judged by the physician as unlikely to be compliant with the study protocol).
* Pregnant or breastfeeding women.
* Patient under legal protection measure.
* Patient is a participating in another research study

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
The stability of the Non-invasive diagnostic test for steatohepatitis (NIS) 4 score and its individual components between the fed and fasting state by the the measurement of the four biomarkers involved in the calculation of NIS4 score | After dinner , 10 hours post-prandial and 12 hours post-prandial

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital la pitié, Paris, France